CLINICAL TRIAL: NCT06639724
Title: A Phase 1b Trial of Perioperative Fostamatinib With Gemcitabine and Nab-paclitaxel in Resectable Pancreatic Cancer
Brief Title: Perioperative Fostamatinib With Gemcitabine and Nab-paclitaxel in Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Hitendra Patel, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810834
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: PDAC; Pancreatic cancer; chemotherapy; Syk kinase inhibitor; Phase 1b; pancreatectomy; biomarkers; tumor microenvironment; non metastatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — fostamatinib; Drug Therapy; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fostamatinib in combination with gemcitabine/nab-paclitaxel (Experimental): Fostamatinib 100 mg will be taken by the study participants orally twice a day for 7 days prior to, and then during chemotherapy with gemcitabine/nab-paclitaxel. These 2 agents will be administered intravenously on days 1, 8, and 15 of each 28-day cycle.
  Interventions: Combination Product: Fostamatinib in combination with chemotherapy (gemcitabine and nab-paclitaxel)

INTERVENTIONS:
Combination Product: Fostamatinib in combination with chemotherapy (gemcitabine and nab-paclitaxel) — Fostamatinib is a Syk kinase inhibitor currently FDA-approved for chronic idiopathic thrombocytopenia purpura but it has not been studied in PDAC. The investigators hypothesize that Syk inhibition reprograms macrophages to an immunostimulatory phenotype in the tumor microenvironment. Thus, Syk inhibition with fostamatinib in combination with chemotherapy could improve outcomes for patients with PDAC while having a favorable safety profile.

SUMMARY:
This is a Phase 1b trial evaluating the combination of Fostamatinib, a Syk kinase inhibitor currently FDA-approved for chronic idiopathic thrombocytopenia purpura (ITP), with the standard of care chemotherapy agents gemcitabine and nab-paclitaxel, for the perioperative treatment of resectable non metastatic pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Although immune checkpoint inhibition has transformed the treatment of some solid malignancies, it has made minimal impact in pancreatic ductal adenocarcinoma (PDAC), which is characterized by a profoundly immunosuppressive microenvironment. Recent published work by the study investigators demonstrated that inhibition of the Syk kinase - alone and in combination with gemcitabine - in preclinical models of PDAC (animal tumor models and human tissues) reprogrammed tumor associated macrophages resulting in enhanced anti-tumor immunity. With this phase Ib study, the investigators aim to expand the preclinical findings to patients with PDAC. This study will evaluate perioperative fostamatinib in combination with standard of care chemotherapy with gemcitabine and nab-paclitaxel. Study participants will receive 4 cycles preoperatively, followed by pancreatic surgical resection and 2 cycles postoperatively. Participants will be followed long term until death or until 2 years after enrollment, whichever occurs first, to evaluate safety and efficacy of perioperative fostamatinib in combination with gemcitabine and nab-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has the ability to understand and willingness to sign a written informed consent.
2. Patient is ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
4. Patient must have surgical consult to verify patient is a surgical candidate within 28 days prior to enrollment.
5. Patient must have resectable primary PDAC based on contrast-enhanced CT or MRI of the chest, abdomen, and pelvis performed no more than 4 weeks before enrollment/baseline. Note that if CT or MRI was performed more than 4 weeks before this visit, imaging needs to be repeated to evaluate eligibility in the study. Resectable primary tumor is defined as:

   1. No involvement of the celiac artery, common hepatic artery, and superior mesenteric artery (and, if present, replaced right hepatic artery).
   2. No involvement, or < 180° interface between tumor and vessel wall, of the portal vein and/or superior mesenteric vein.
   3. Patent portal vein/splenic vein confluence.
   4. No evidence of metastatic disease.
   5. Lymphadenopathy (defined as nodes measuring > 1cm in short axis) outside the surgical basin (i.e., para- aortic, peri-caval, celiac axis, or distant nodes) is considered M1 disease and makes the patient ineligible. If, however, such nodes are biopsied and are negative, then enrollment can be considered after review with the study principal investigator (PI) and/or co-investigator.
   6. For tumors of the body and tail of the pancreas, involvement of the splenic artery and vein of any degree is considered resectable disease.
6. Patient has adequate organ function as defined below:

   1. Absolute Neutrophil Count ≥ 1.5 x 10^9/L
   2. Platelet count ≥ 100 x 10^9/L.
   3. Hemoglobin ≥ 9.0 g/dL
   4. aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SPGT) ≤ 2.5 X institutional upper limit of normal (ULN)
   5. Total Bilirubin ≤ 1.5 x institutional ULN or ≤3 × institutional ULN in Gilbert's Ds
   6. Serum creatinine ≤ 2 x institutional ULN
7. For subjects able to become pregnant: use of highly effective contraception for at least 2 weeks prior to enrollment and agreement to use such a method during study participation.
8. For subjects able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner during study participation.

Exclusion Criteria:

1. Any prior treatment for PDAC.
2. Recurrent or metastatic PDAC.
3. Peripheral neuropathy > grade 2
4. Received an investigational agent within 28 days prior to the first dose of study drug.
5. History of Hepatitis B (defined as Hepatitis B surface antigen, HBsAg, reactive) or known active Hepatitis C virus (HCV) (defined as HCV RNA - qualitative - is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority. (Individuals who are hepatitis C antibody positive may be enrolled if negative viral load confirmed).
6. Active infection requiring systemic therapy.
7. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. History of receiving a solid organ transplant or allogeneic bone marrow transplant.
9. Major surgical procedure within 28 days prior to the first dose of study drug.
10. Unable or unwilling to withhold or discontinue any prohibited or restricted medications/procedures for the specified windows during the study.
11. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Surgical delay | 6 weeks from the last pre-operative treatment cycle
  Number and percentage of participants who experience surgical delay, as measured by the proportion of enrolled participants for whom pancreatic resection cannot be performed within 6 weeks of the last pre-operative treatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lowy, MD, Study Chair — UCSD
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available

REFERENCES:
- [Background] Rohila D, Park IH, Pham TV, Weitz J, Hurtado de Mendoza T, Madheswaran S, Ishfaq M, Beaman C, Tapia E, Sun S, Patel J, Tamayo P, Lowy AM, Joshi S. Syk Inhibition Reprograms Tumor-Associated Macrophages and Overcomes Gemcitabine-Induced Immunosuppression in Pancreatic Ductal Adenocarcinoma. Cancer Res. 2023 Aug 15;83(16):2675-2689. doi: 10.1158/0008-5472.CAN-22-3645. PMID 37306759